CLINICAL TRIAL: NCT06106971
Title: Balloon-occluded Retrograde Transvenous Obliteration Versus Endoscopic Tissue Glue Injection in the Prevention of Recurrent Gastric Variceal Bleeding
Brief Title: Balloon-occluded Retrograde Transvenous Obliteration for Gastric Variceal Rebleeding
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Wen-Chi Chen, Doctor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS18-CT6-12
Record Dates: First submitted 2023-10-17; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Gastric Varices Bleeding; Liver Decompensation
Keywords: gastric varices bleeding; cyanoacrylate; balloon-occluded retrograde transvenous obliteration; liver decompensation; cirrhosis
MeSH Terms: conditions — Hepatic Insufficiency; Fibrosis | interventions — Sodium Tetradecyl Sulfate; Cyanoacrylates

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon-occluded retrograde transvenous obliteration (Experimental): Information of drug:
  3% sodium tetradecyl sulfate injection Name: Fibro-vein injection Manufacturer: STD Pharmaceutical Products Ltd.
  Interventions: Drug: Sodium tetradecyl sulfate
- Endoscopic cyanoacrylate injection (Active Comparator): Information of drug:
  N-butyl-2-cyanoacrylate Name: Histoacryl blue Manufacturer: Braun, Melsungen, Germany
  Interventions: Drug: Cyanoacrylate

INTERVENTIONS:
Drug: Sodium tetradecyl sulfate — Subjects receive sodium tetradecyl sulfate via balloon-occluded retrograde transvenous obliteration at 3 to 5 days after initial hemostasis of acute gastric variceal bleeding.
  Arms: Balloon-occluded retrograde transvenous obliteration
Drug: Cyanoacrylate — Subjects receive endoscopic cyanoacrylate injection at 3 to 5 days after initial hemostasis of acute gastric variceal bleeding then receive repeated endoscopic cyanoacrylate injection at 1-month intervals until obliteration of gastric varices.
  Arms: Endoscopic cyanoacrylate injection

SUMMARY:
The goal of this randomized controlled trial is to compare the rebleeding rate in cirhotic patients with gastric variceal bleeding receiving balloon-occluded retrograde transvenous obliteration and endoscopic tissue glue injection. The main questions it aims to answer are:

* Recurrent gastric variceal bleeding
* Further decompensation of liver cirrhosis

Participants will receive balloon-occluded retrograde transvenous obliteration and endoscopic tissue glue injection. Researchers will compare balloon-occluded retrograde transvenous obliteration and endoscopic tissue glue injection to see if the rebleeding rate associated with balloon-occluded retrograde transvenous obliteration is lower than that associated with endoscopic tissue glue injection.

DETAILED DESCRIPTION:
Variceal bleeding is a severe complication of portal hypertension. Gastric variceal bleeding (GVB) is more severe than bleeding from esophageal varices. Gastric varices also have a higher risk of rebleeding than esophageal varices. Previous studies showed that endoscopic injection of cyanoacrylate was superior to endoscopic variceal ligation in the management of gastric variceal bleeding. Another study showed that transjugular intrahepatic portosystemic shunt had a lower rebleeding rate than endoscopic cyanoacrylate injection. However, transjugular intrahepatic portosystemic shunt (TIPS) is more invasive and carries a risk of development of hepatic encephalopathy and is usually preserved for uncontrolled variceal bleeding. Therefore, endoscopic cyanoacrylate injection is recommended as the treatment of choice for GVB. Balloon-occluded retrograde transvenous obliteration (BRTO) is a new therapy for gastric variceal bleeding. However, BRTO is associated with increased portal pressure and worsening of ascites, hepatohydrothorax, and esophageal varices. There are only a few retrospective studies comparing BRTO and endoscopic cyanoacrylate injection in the prevention of recurrent gastric variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

* age more than 20 years
* a history of liver cirrhosis
* acute GOV2 or IGV1 bleeding

Exclusion Criteria:

* previous treatment for gastric varices, including endoscopic therapy, transjugular intrahepatic portosystemic shunt, or shunt surgery
* hepatocellular carcinoma or other malignancy
* stroke, uremia, or active sepsis
* serum total bilirubin >10 mg/dL
* grade III/IV hepatic encephalopathy
* refractory ascites
* uncontrolled index bleeding
* pregnancy
* severe heart failure (NYHA Fc III/IV)
* allergy to cyanoacrylate, lipiodol, iodine, or sodium tetradecyl sulfate
* absence of gastrorenal shunt

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
recurrent gastric variceal bleeding | From date of randomization until the date of first documented recurrent gastric variceal bleeding or date of death from any cause, whichever comes first, assessed up to 100 months
  recurrent gastric variceal bleeding after interventions
further liver decompensation | From date of randomization until the date of first documented further liver decompensation or date of death from any cause, whichever comes first, assessed up to 100 months
  further liver decompensation after intervensions

SECONDARY OUTCOMES:
recurrent upper gastrointestinal bleeding | From date of randomization until the date of first documented recurrent upper gastrointestinal bleeding or date of death from any cause, whichever comes first, assessed up to 100 months
  recurrent upper gastrointestinal bleeding after interventions
mortality or liver transplantation | From date of randomization until the date of documented liver transplantation or date of death from any cause, whichever comes first, assessed up to 100 months
  mortality or liver transplantation after intervensions

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chi Chen, M.D, Principal Investigator — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared 12 months after article publication.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 12 months after article publication and the data will be made accessible for up to 24 months.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan and execution of a Data Sharing Agreement. For more information or to submit a request, please contact wcchen@vghks.gov.tw.

REFERENCES:
- [Background] Ryan BM, Stockbrugger RW, Ryan JM. A pathophysiologic, gastroenterologic, and radiologic approach to the management of gastric varices. Gastroenterology. 2004 Apr;126(4):1175-89. doi: 10.1053/j.gastro.2004.01.058. PMID 15057756
- [Background] Sarin SK, Lahoti D, Saxena SP, Murthy NS, Makwana UK. Prevalence, classification and natural history of gastric varices: a long-term follow-up study in 568 portal hypertension patients. Hepatology. 1992 Dec;16(6):1343-9. doi: 10.1002/hep.1840160607. PMID 1446890
- [Background] Rockey DC. Management of gastric varices. Gastroenterology. 2001 Jun;120(7):1875-6; discussion 1876-7. doi: 10.1053/s0016-5085(01)70197-7. No abstract available. PMID 11375970
- [Background] Tripathi D, Therapondos G, Jackson E, Redhead DN, Hayes PC. The role of the transjugular intrahepatic portosystemic stent shunt (TIPSS) in the management of bleeding gastric varices: clinical and haemodynamic correlations. Gut. 2002 Aug;51(2):270-4. doi: 10.1136/gut.51.2.270. PMID 12117893
- [Background] Park JK, Saab S, Kee ST, Busuttil RW, Kim HJ, Durazo F, Cho SK, Lee EW. Balloon-Occluded Retrograde Transvenous Obliteration (BRTO) for Treatment of Gastric Varices: Review and Meta-Analysis. Dig Dis Sci. 2015 Jun;60(6):1543-53. doi: 10.1007/s10620-014-3485-8. Epub 2014 Dec 18. PMID 25519690
- [Background] Tan PC, Hou MC, Lin HC, Liu TT, Lee FY, Chang FY, Lee SD. A randomized trial of endoscopic treatment of acute gastric variceal hemorrhage: N-butyl-2-cyanoacrylate injection versus band ligation. Hepatology. 2006 Apr;43(4):690-7. doi: 10.1002/hep.21145. PMID 16557539